CLINICAL TRIAL: NCT05786625
Title: Assessment of the Safety and Performance of the AB1 Electrosurgical System for Bronchoscopic Microwave Ablation of Lung Tissue
Brief Title: Bronchoscopic Microwave Ablation of Lung Tissue
Acronym: AB1MALT
Status: Active, not recruiting | Type: Observational
Sponsor: Creo Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-AB1-950
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Neoplasms; Bronchoscopy; Ablation; Microwave
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Microwave ablation: Patients with a single or multiple soft tissue lung lesions that is medically inoperable or for which the patient has declined surgical resection.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Bronchoscopy and microwave ablation of lung nodule

SUMMARY:
The primary purpose of this study is to evaluate the safety and feasibility of the Creo Medical MicroBlate™ Flex AB1 instrument used with the AB1 electrosurgical system in patients undergoing bronchoscopic microwave ablation of peripheral lung nodules.

DETAILED DESCRIPTION:
This is a post-market, prospective, single-arm, multicentre, non-randomized, observational study which will enrol up to 35 subjects in total (plus replacements) at up to 6 clinical investigation sites in Europe and potentially 1 site in the US.

Prospective patients must have a suitable soft tissue lung lesion and be candidates for an elective endobronchial navigation and microwave ablation procedure performed bronchoscopically. After being informed about the study and potential risks, all patients giving their written informed consent will undergo a screening visit to determine eligibility for study entry. Patients who meet the eligibility requirements will undergo a pre-procedural assessment, a bronchoscopy procedure that includes ablation treatment with MicroBlate™ Flex AB1, a post-procedural assessment and 6 follow-up visits at, 7 days (by phone call or in person), 31-45 days, 3 months, 6 months, 9 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

The participant may enter the study if ALL of the following apply:

The patient:

1. Has signed the informed consent form
2. Are ≥ 18 years old
3. Has lung lesion(s)/nodule(s) which are histologically confirmed or highly suspicious for cancer and is a candidate for bronchoscopic microwave ablation (as determined by a multi-disciplinary team (MDT) or tumour board).
4. Has a medically inoperable soft tissue lung lesion(s) ≤ 20 mm (suspected or confirmed malignancy), or patient has elected not to have surgery / alternative therapy.
5. Patient is a candidate for bronchoscopy under general anaesthesia.
6. Subject is willing and able to comply with the study protocol requirements.
7. Are assigned an ASA (American Society of Anaesthesiologists) score of ≤ 3 or the patient is deemed fit for general anaesthesia.

Exclusion Criteria:

The participant may not be enrolled in the study if ANY of the following apply:

For patients undergoing procedures employing robotic-assisted bronchoscopy:

1. a. Target nodule(s) are within 10mm of the trachea, right and left main bronchus, aorta, central pulmonary arteries, heart, oesophagus, spinal cord, phrenic & laryngeal nerves.

Note: Exclusion Criteria 1a is UK-specific.

For patients undergoing procedures without the use of robotic-assisted bronchoscopy (manual procedures):

1. b. Target nodule(s) are within the International Association for the Study of Lung Cancer (IASLC) "Central Zone" (including bronchial tree, major vessels, heart, oesophagus, spinal cord and phrenic and laryngeal nerves), or are <10 mm from the pleura.
2. Are assigned status 4 via ECOG (Eastern Cooperative Oncology Group) classification.
3. Are pregnant or breast feeding, as determined by standard site practices.
4. Have participated in an investigational drug or device research study within 30 days of enrolment that would interfere with this study.
5. Are scheduled for concurrent interventional procedure for the target soft tissue lesion.
6. Have a physical or psychological condition or other factor(s) that would impair study participation, or jeopardise the safety or welfare of the subject.
7. Have an expected survival less than 6 months.
8. Have patients with bleeding diathesis, uncorrectable coagulopathy or platelet count ≤ 100 x 10⁹ /L.
9. Have an implantable devices, including pacemakers or other electronic implants.
10. Have known pulmonary hypertension (PASP [pulmonary artery systolic pressure] > 50mmHg).
11. Who are currently prescribed anticoagulants, clopidogrel or other platelet aggregation inhibitors which cannot be stopped or temporarily withheld.
12. Any patient with clinically significant interstitial lung disease in the zone of planned ablation.

    Note: Exclusion Criteria 12 is NL-specific.
13. Patient has nodal disease confirmed through invasive or image-based staging. Note: if nodal disease is suspected or detected during the staging procedure conducted prior to use of the investigational device during the study procedure, the subject will be excluded.
14. Subject had a prior pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the proposed study must have a suitable soft tissue lung lesion and be candidates for an elective endobronchial navigation and microwave ablation procedure performed bronchoscopically. Patients without a histologically confirmed diagnosis of cancer may be enrolled if a multi-disciplinary board deems that it is highly likely that their lung lesion is a malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Performance (Efficacy) Endpoint | Up to day 30 patient visit.
  Initial technical success, defined as successful bronchoscopic access by the AB1 instrument of the target tissue, delivery of the scheduled microwave energy to the target tissue and confirmed ablation as evidenced by assessment of CT.
  The criterion for meeting the Performance (efficacy) endpoint excludes study system malfunctions.
Primary Safety Endpoint | Up to 30 days after the ablation procedure.
  Identification of serious device-related adverse events related to the use of the AB1 system up to 30 days after the ablation procedure (number and nature of serious adverse events, both device- and procedure- related, will be identified) including, but not limited to:
  * Moderate bleeding (intervention required such as use of balloon tamponade or Surgicel) or severe bleeding (prolonged monitoring necessary or fatal bleeding)
  * Pneumothorax
  * Failure of extubation
  * ICU admission for respiratory failure within 30 days
  * Death within 30 days.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | Up to 12 months post ablation.
  Identification of all device-related, procedure related and other adverse events related to bronchoscopic microwave ablation interventions using the AB1 system.
Secondary Effectiveness Outcomes - Rate of tumor recurrence | Up to 12 months
  Rate of recurrence at all time points as determined by the multidisciplinary team (MDT) or tumour board.
Secondary Effectiveness Outcomes - European Organization for Research and Treatment of Cancer Quality of life questionnaire - Cancer (EORTC QLQ-C) | Up to 12 months
  Patients will rate their responses from 1 to 4 on a Likert Scale (1 being "not at all" and 4 being "very much").
Secondary Effectiveness Outcomes - EQ-5D-5L health-related quality of life questionnaire | Up to 12 months
  Patients complete the 5 level descriptive system relating to 5 dimensions of health and the EQ visual analogue scale from 0 to 100 (where 0 means the worst health you can imagine and 100 means the best health you can imagine).
Secondary Effectiveness Outcomes - Patient-reported pain rating on a visual analogue scale | Up to 45 days post-ablation
  Patients will rate their pain on a visual analogue scale from 0 to 10 (where 0 is no pain and 10 is the most severe pain).
Secondary Effectiveness Outcomes - Assessment/visualization/quantification of the dimensions of the ablated tissue | Up to 12 months
  Dimensions of the ablated tissue to confirm, correct or add to the IFU-reported relationship between AB1 ablation time and dimensions and volume of the ablated tissue, per pre-specified target.
Secondary Effectiveness Outcomes - Procedural Time | Up to 1 day post ablation procedure.
  Procedural time to be captured in the electronic case report form (eCRF).
Secondary Effectiveness Outcomes - Assessment of ease of system use (clinician questionnaires) | Up to 1 day post ablation procedure.
  Questionnaires to be completed by clinicians, rating their responses on a Likert scale of 1 to 7, with 1 being "extremely easy" and 7 being "extremely difficult".

CONTACTS AND LOCATIONS:
Overall Officials: Pallav L Shah, MD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (2):
- Amsterdam University Medical Centres, Location AMC, Meibergdreef 9, Amsterdam, Netherlands
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Single site